CLINICAL TRIAL: NCT07059117
Title: High Versus Low Versus Optimal Umami Taste Intensity in a Risotto Mixed Meal With Comparable Palatability on ad Libitum Meal Intake
Brief Title: Umami Taste Intensity and ad Libitum Meal Intake
Acronym: RiceSort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Principal Investigator, Ciaran Forde, Prof. Dr., Wageningen University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NL51747.081.14
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-06

CONDITIONS: Taste Sensitivity; Umami Taste Perception; Food Intake Regulation; Hedonic Function; Palatability
Keywords: umami; savoury; ad libitum; taste intensity; palatability; food intake; hedonic mapping; MSG

STUDY DESIGN:
Intervention Model Description: Complete block randomized cross-over design.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low umami intensity (Experimental): The low umami intensity meal will have a taste intensity corresponding with the MSG concentration in the sample rated 1.85 units to the left on the Visual Analogue Scale (VAS) during the first test session in which umami taste preferences per individual will be assessed by hedonic mapping.
  Interventions: Other: Hedonic mapping; Other: Ad libitum risotto test meal
- High umami intensity (Experimental): The high umami intensity meal will have a taste intensity corresponding with the MSG concentration in the sample rated 1.85 units to right left on the Visual Analogue Scale (VAS) during the first test session in which umami taste preferences per individual will be assessed by hedonic mapping.
  Interventions: Other: Hedonic mapping; Other: Ad libitum risotto test meal
- Optimum umami taste intensity (Experimental): The optimum umami intensity meal will have a taste intensity corresponding with the MSG concentration in the sample rated closest to the 'Just right' point on the Visual Analogue Scale (VAS) during the first test session in which umami taste preferences per individual will be assessed by hedonic mapping.
  Interventions: Other: Hedonic mapping; Other: Ad libitum risotto test meal

INTERVENTIONS:
Other: Hedonic mapping — During the first session, participants will be presented with risotto samples differing in MSG content and thus umami taste intensity, assigned based on Booth's method (Booth et al., 1983). Based on these individual ratings, umami taste intensities of the ad libitum test meals will be calculated per participant.
Other: Ad libitum risotto test meal — During the ad libitum test meal, participants will be presented with 800 grams of risotto with either high-, low-, or optimum umami taste intensity.

SUMMARY:
Background Sweet and salty tastes can influence food intake {Sørensen, 2003 #40}. Increased intensity of these tastes has been shown to decrease food intake and increase satiation compared to the less intense taste, independent of palatability {Bolhuis, 2010 #245;Bolhuis, 2011 #251;Chung, 2007 #253;Lucas, 1987 #258;Vickers, 1998 #252;Vickers, 1998 #249;Vickers, 2001 #246;Yeomans, 1998 #244}. Umami taste intensity has been shown to reduce subsequent food intake {Masic, 2014 #7}, especially when paired with protein content in foods {Masic, 2014 #6}. Taste can be related with nutrient content of the diet, with sweet foods having carbohydrates, salty foods containing sodium, and umami foods containing protein {Teo, 2018 #37}.

However, no study has yet investigated the impact of umami and food intake, using the approach of similar palatability and differing taste intensity levels {Forde, 2016 #254}. Given its relationship with nutrient signaling, it is important to explore the relationship between umami intensity and satiation. Therefore, this study aims to compare ad libitum food intake of two levels with similar palatability and differing umami taste intensities (high and low) to food intake from a meal with optimum taste intensity.

Methods Test session 1 Determine individual's most preferred level of umami taste in 10 risotto samples, use Booth's method {Booth, 1983 #247}. Samples will contain a fixed level of salt, and MSG concentrations ranging from 0.2-1.2 w/w%, based on the optimal amount of MSG added to enhance taste to be 0.1-0.8 w/w% {Wijayasekara, 2017 #70}. Per individual, samples that are closest to those situated at -3.5 and +3.5 from the optimum (at 7) will be selected (figure 1).

Healthy, normal weight participants will be included. Previous studies have applied this method in sweet and salty tastes with 15-59 participants {Bolhuis, 2010 #245;Bolhuis, 2011 #251;Bolhuis, 2012 #255;Vickers, 1998 #252;Vickers, 1998 #249;Vickers, 2001 #246}.

Test session 2, 3 and

In a randomized cross-over design, participants will receive the optimum, high and low MSG risotto. The following will be measured:

* Test meal consumption (primary outcome);
* Liking before meal;
* Liking after meal;
* Water consumption;
* Taste intensity ratings of the meal;
* Habitual dietary taste exposure (tasteFFQ).

Subjects will be asked to eat a similar breakfast and to not consume anything between breakfast and lunch session. They will also be asked to refrain from eating for one hour after the test session. Participants will be asked to fill in the tasteFFQ, to investigate the link between dietary taste patterns and hedonic umami taste ratings.

Data will be analyzed using Rstudio. First, normality will be assessed, and data will be normalized if needed. Difference in food intake in grams between the three intensities will be compared using ANOVA. A post-hoc test will be applied if statistical outcomes are significant. Categorical variables will be compared using Chi-square test.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported healthy;
* BMI between 18.5 and 25 kg/m2;
* Age between 18 and 55 years old;
* Able to visit the research facilities on the Wageningen campus for hedonic mapping (once) and for the risotto lunch meal (three times);
* Able to provide informed consent.

Exclusion Criteria:

* Diagnosed with smell- or taste disorder(s);
* Use of medication that could influence taste ability and/or food intake behaviour;
* Food allergy or intolerance to any of the ingredients used in the ad libitum test meal;
* Consumption of more than 14 (women) or 21 (men) glasses of alcohol per week;
* Student or personnel of the Health Research Unit at Wageningen University

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2025-04-12 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
Difference in food intake from ad libitum test meal between taste intensity conditions | Test session 2, 3, and 4 (week 2, 3 and 4)
  Difference in food intake in volume (grams) from the ad libitum test meal between the three (high-, low- and optimum) umami taste intensities.

SECONDARY OUTCOMES:
Difference in liking before meal between taste intensity conditions | Test session 2, 3, and 4 (week 2, 3 and 4)
  Difference in test meal liking, measured on a Visual Analogue Scale, 0-100 (0 representing not liking at all, 100 representing like very much) between the three (high-, low- and optimum) umami taste intensities.
Difference in liking after meal between taste intensity conditions | Test session 2, 3, and 4 (week 2, 3 and 4)
  Difference in test meal liking, measured on a Visual Analogue Scale, 0-100 (0 representing not liking at all, 100 representing like very much) between the three (high-, low- and optimum) umami taste intensities.
Difference in umami taste intensity ratings of the ad libitum test meal between taste intensity conditions | Test session 2, 3, and 4 (week 2, 3 and 4)
  Difference in taste intensity ratings of the ad libitum test meal, measured on a Visual Analogue Scale, 0-100 (0 representing no umami taste at all, 100 representing very intense umami taste) between the three (high-, low- and optimum) umami taste intensities.
Difference in water consumption during the ad libitum test meal between taste intensity conditions | Test session 2, 3, and 4 (week 2, 3 and 4)
  Difference in water consumption in volume (grams) from the ad libitum test meal between the three (high-, low- and optimum) umami taste intensities.
Difference in reported appetite and fullness ratings between the three conditions | Test session 2, 3, and 4 (week 2, 3 and 4)
  Before and after the ad libitum test meals, appetite and fullness ratings of participants, measured on a Visual Analogue Scale, 0-100 (0 representing not at all, 100 representing very much). Differences of these rating between umami taste intensity conditions (low-, high- and optimum umami taste intensity) will be assessed.
Habitual taste exposure | The month prior to the first ad libitum test meal (session 2).
  Habitual taste exposure will be measured with a food frequency questionnaire (tasteFFQ) specifically designed to assess relative food intake based on taste cluster. Individual optimum umami intensity will be compared to habitual dietary taste exposure to the salt, umami and fat taste cluster, as well as to the intake of umami tasting food items.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Mars, PhD, Principal Investigator — Wageningen University; Ciaran Forde, PhD, Study Chair — Wageningen University
Locations (1):
- Department of Human Nutrition, Wageningen University, Wageningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Individual study participant data will be shared after anonymization upon study publication in an open data repository (e.g. DANS or Yoda).

REFERENCES:
- [Background] Jayasena DD, Kang T, Wijayasekara KN, Jo C. Innovative Application of Cold Plasma Technology in Meat and Its Products. Food Sci Anim Resour. 2023 Nov;43(6):1087-1110. doi: 10.5851/kosfa.2023.e31. Epub 2023 Nov 1. PMID 37969327
- [Background] Forde, C. G. (2016). Flavor perception and satiation. In Flavor (pp. 251-276). Woodhead Publishing.
- [Background] Masic U, Yeomans MR. Monosodium glutamate delivered in a protein-rich soup improves subsequent energy compensation. J Nutr Sci. 2014 Aug 13;3:e15. doi: 10.1017/jns.2014.15. eCollection 2014. PMID 25191607
- [Background] Bolhuis DP, Lakemond CM, de Wijk RA, Luning PA, de Graaf C. Effect of salt intensity in soup on ad libitum intake and on subsequent food choice. Appetite. 2012 Feb;58(1):48-55. doi: 10.1016/j.appet.2011.09.001. Epub 2011 Sep 29. PMID 21986190
- [Background] Bolhuis DP, Lakemond CM, de Wijk RA, Luning PA, Graaf Cd. Both longer oral sensory exposure to and higher intensity of saltiness decrease ad libitum food intake in healthy normal-weight men. J Nutr. 2011 Dec;141(12):2242-8. doi: 10.3945/jn.111.143867. Epub 2011 Nov 2. PMID 22049294
- [Background] Bolhuis DP, Lakemond CM, de Wijk RA, Luning PA, de Graaf C. Effect of salt intensity on ad libitum intake of tomato soup similar in palatability and on salt preference after consumption. Chem Senses. 2010 Nov;35(9):789-99. doi: 10.1093/chemse/bjq077. Epub 2010 Aug 12. PMID 20705808
- [Background] Sorensen LB, Moller P, Flint A, Martens M, Raben A. Effect of sensory perception of foods on appetite and food intake: a review of studies on humans. Int J Obes Relat Metab Disord. 2003 Oct;27(10):1152-66. doi: 10.1038/sj.ijo.0802391. PMID 14513063
- [Background] Masic U, Yeomans MR. Umami flavor enhances appetite but also increases satiety. Am J Clin Nutr. 2014 Aug;100(2):532-8. doi: 10.3945/ajcn.113.080929. Epub 2014 Jun 18. PMID 24944058